CLINICAL TRIAL: NCT03435848
Title: A Phase 2b Open-Label, Single Arm, Multi-Center Study to Assess the Efficacy and Safety of BST-236 as a Single Agent in Adults With Newly-Diagnosed Acute Myeloid Leukemia (AML), Not Eligible for Standard Induction Therapy
Brief Title: Efficacy and Safety of BST-236 in Newly Diagnosed Acute Myeloid Leukemia Patients, Unfit for Standard Induction Therapy
Acronym: ELPIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioSight Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BST002
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Unfit for standard induction therapy; Cytarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BST-236 (Experimental): BST-236 Intravenous, 4.5 g/m2/d or 2.5 g/m2/d, for 6 days
  Interventions: Drug: BST-236

INTERVENTIONS:
Drug: BST-236 — 1 to 4 courses

SUMMARY:
The purpose of this study is to assesses the benefit, safety, and pharmacokinetics (PK) of BST-236 in patients with newly-diagnosed Acute Myeloid Leukemia (AML) who are not eligible for standard induction chemotherapy due to advanced age or comorbidities. The Complete Remission (CR) rate following treatment with BST-236 will be compared to the CR rate reported in historical data in a similar population.

DETAILED DESCRIPTION:
BST-236 is a cytarabine pro drug designed to release cytarabine inside the target cells with reduced systemic exposure to free cytarabine. As such, BST-236 may enable delivery of high doses of cytarabine to medically-unfit or older adults who otherwise cannot be treated with standard cytarabine therapy. This study aims to validate this hypothesis.

The study is an open-label, single arm, single agent, multi-center study in adults with newly diagnosed AML who are unfit for standard therapy. The patients will receive up to 4 courses of six-days treatment with intravenous BST-236; 1 or 2 induction courses followed by 1 to 2 consolidation courses. The study participation will be 52 weeks including treatment and follow-up periods. An additional 1 year post study follow-up for the evaluation of survival is optional.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥18 years of age
2. AML according to the 2016 revision to the World Health Organization (WHO) classification of myeloid neoplasms and acute leukemia: ≥20% blasts in peripheral blood or marrow

   1. de-novo AML or
   2. AML secondary to MDS or
   3. AML secondary to exposure to potentially leukemogenic therapies or agents (e.g. radiation therapy, alkylating agents, topoisomerase II inhibitors) with the primary malignancy in remission for at least 2 years
3. Not eligible for standard induction chemotherapy;

   1. Age ≥75 years or
   2. Age ≥18 years with at least one of the following comorbidities:

   i. Clinically significant heart or lung comorbidities, as reflected by at least one of:
   * Left ventricular ejection fraction (LVEF) ≤50%
   * Lung diffusing capacity for carbon monoxide (DLCO) ≤65% of expected
   * Forced expiratory volume in 1 second (FEV1) ≤65% of expected ii. Chronic stable angina or congestive heart failure controlled with medication iii. Other contraindication(s) to anthracycline therapy (must be documented) iv. Other comorbidity that the Investigator judges as incompatible with intensive remission induction chemotherapy, which must be documented
4. Creatinine clearance (estimated by the Cockroft-Gault (C-G) or measured by 24 hours urine collection) ≥45 mL/min
5. Liver enzymes (aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤2.5 times the upper limits of normal (ULN)
6. Total bilirubin ≤1.5 x ULN unless due to known history of Gilbert's disease
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 at screening
8. Prepared and able to give written (signed and dated) informed consent, which includes compliance with study requirements and restrictions prior to admission to the study
9. Women of reproductive potential must have a negative serum pregnancy test within 48 hours of the first day of any BST-236 treatment course
10. Women or men of reproductive potential must use (or have his/her partner use) two forms of effective birth control methods starting from 1 month prior to screening and until 3 months following the last BST-236 administration day (acceptable methods of birth control in this study include: surgical sterilization, intrauterine devices, oral contraceptives, contraceptive patch, long-acting injectable contraceptives, partner's vasectomy, or double-barrier method condom or diaphragm with spermicide)
11. Patient must voluntarily sign and date an ICF, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures
12. Patient must be able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Patient has relapsed or refractory AML
2. Patient has acute promyelocytic leukemia
3. Any previous treatment for AML (except for hydroxyurea or up to one treatment course with hypomethylating agents (HMA))
4. Patient has history of myeloproliferative neoplasm (MPN) including myelofibrosis, essential thrombocythemia, polycythemia vera, chronic myeloid leukemia (CML) with or without BCR-ABL1 translocation and AML with BCR-ABL1 translocation
5. Previous use (prior to study initiation) of drugs containing cytarabine as an active ingredient
6. Use of any HMA for the treatment of MDS within 30 days of study Day 1
7. Participation in a previous clinical trial and/or use of an investigational drug within 90 days or at least 5 half-lives of tested drug (whichever is longer) of initial screening assessment
8. Peripheral White Blood Cell (WBC) count >30,000 /µL in the 48 hours prior to first BST-236 dose administration. Hydroxyurea administration or leukapheresis is permitted to meet this criterion
9. Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment)
10. Any medical or surgical condition, presence of laboratory abnormalities or psychiatric illness that may preclude safe and complete study participation based on the Investigator's judgment
11. Diagnosis of malignant disease within the previous 12 months (excluding basal cell carcinoma of the skin without complications, "in-situ" carcinoma, or other local malignancy excised or irradiated with a high probability of cure and not treated with chemotherapy)
12. Active malignant disease other than AML
13. Leptomeningeal/central nervous system involvement of AML
14. Myeloid sarcoma as a sole manifestation of AML
15. Surgical procedure, excluding central venous catheter placement or other minor procedures (e.g. skin biopsy) in the 14 days prior to BST-236 administration
16. Unstable angina, significant cardiac arrhythmia, or New York Heart Association (NYHA) class 4 congestive heart failure
17. Shortness of breath requiring continuous oxygen treatment for at least 15 hours per day in chronically hypoxemic patients
18. History of allergic reactions attributed to compounds of similar chemical composition as BST-236 and/or cytarabine
19. Life expectancy shorter than 3 months attributed to any known medical condition other than AML
20. Active/chronic Hepatitis B Virus (HBV) infection (based on positive surface antigen (HBsAg)), Hepatitis C Virus (HCV) infection (HCV) (based on positive HCV antibody (Ab)), or Human Immunodeficiency Virus (HIV)-1 or HIV-2 (based on positive HIV antibody)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Complete Remission | Day 28-35 of induction/re induction course
  as BM blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC >1.0x 109/L (1,000/μL); platelet count >100 x 109/L (100,000/μL)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (11):
  - Augusta University Georgia Cancer Center, Augusta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Franciscan Physician Network Oncology and Hematology Specialists, Indianapolis, Indiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center New York, New York, New York
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute, Columbus, Ohio
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - Baylor Scott & White Research Institute Dallas Texas, Dallas, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
- Israel (5):
  - Soroka University Medical Center, Beersheba
  - Rambam medical center hematology department, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Altman JK, Zuckerman T, Koprivnikar J, McCloskey J, Kota V, Keng M, Frankfurt O, Abaza Y, Bixby DL, Emadi A, Burch M, Bhatnagar B, Luger SM, Percival ME, Wolach O, Craig M, Ganzel C, Roboz G, Levi I, Gourevitch A, Flaishon L, Tessler S, Blumberg C, Gengrinovitch S, Ben Yakar R, Rowe JM. Aspacytarabine for the treatment of patients with AML unfit for intensive chemotherapy: a phase 2 study. Blood Adv. 2023 Dec 26;7(24):7494-7500. doi: 10.1182/bloodadvances.2023010943. PMID 37903324